CLINICAL TRIAL: NCT02541422
Title: Use of NAC in Alleviation of Hangover Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's Hospital and Health Network, Pennsylvania (Other)
Responsible Party: Principal Investigator, Holly Stankewicz, D.O., Attending physician and faculty emergency medicine residency, St. Luke's Hospital and Health Network, Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SLHN 2015-27
Record Dates: First submitted 2015-09-01; First posted 2015-09-04 (Estimated); Results first posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2017-09

CONDITIONS: Hangover Symptoms, NAC
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NAC group (Active Comparator): Patients receiving NAC after drinking to breathalyzer value 0.1
  Interventions: Dietary Supplement: N Acetyl Cysteine
- Placebo group (Placebo Comparator): Patients receiving placebo after drinking to breathalyzer value 0.1
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: N Acetyl Cysteine
  Other Names: NAC
  Arms: NAC group
Other: placebo
  Arms: Placebo group

SUMMARY:
This will be a double-blinded study involving healthy non-alcoholic (self-reported) volunteers over the age of 21 to consume beer on hospital property in a safe environment to ensure immediate availability to medical attention and to security if needed. Volunteers will be recruited from residency programs, hospital employees, emergency medical personnel, and friends of study investigators. The volunteers will drink to a BAC of 0.1 as checked with a breathalyzer. They will wear a tag around their neck with their study number, which will be hole-punched with every beer consumed, which will be collected at the end of the night for an accurate count of beers consumed per person. They however will not be forced to drink anymore if they are uncomfortable with the amount of alcohol they are consuming and can withdraw from the study at any time. All participants will be required to be driven home by a sober driver once the participant's BAT is 0.02 or less. At the end of the night, the volunteer will be breathalyzed to determine BAC, and given 1 capsule per 3 drinks consumed of either 600 mg N-Acetyl-L-Cysteine or placebo capsules. In the morning, each participate will fill out a Hangover Symptom Score questionnaire, evaluating each hangover symptom on a 0 - 4 point Hangover Symptom Severity scale. A random number generator will be used to determine Placebo or NAC first, then the participant will be given the other treatment at their subsequent encounter. The study will be conducted over the series of many months, and data can be analyzed by self-control comparing the participant's hangover symptom severity as determined by the hangover symptom scale data when using NAC compared to placebo. The data will be analyzed using the numerical values of each category for hangover classification and compare the placebo data to the control data.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers over age 21 years

Exclusion Criteria:

* Volunteers will be excluded from the study if they suffer from any of the following conditions:
* Alcoholism,
* Pregnancy,
* Reactive Airway Disease,
* Diabetes,
* Kidney or bladder stones,
* Kidney disease,
* Liver disease,
* Stomach ulcer,
* Organ transplant patients,
* Dialysis patients,
* and patients with alcohol, egg, milk or wheat allergies.

Volunteers taking the following medications will not be able to participate:

* activated charcoal,
* ampicillin,
* carbamazepine,
* cephaloridine,
* cloxacillin,
* methicillin,
* nitroglycerine,
* oxacillin,
* penicillin G,
* or quinacillin.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly A Stankewicz, D.O., Principal Investigator — St. Luke's Hospital and Health Network, Pennsylvania
Locations (1):
- St. Luke's Hospital, Bethlehem, Pennsylvania, United States

REFERENCES:
- [Result] Swift R, Davidson D. Alcohol hangover: mechanisms and mediators. Alcohol Health Res World. 1998;22(1):54-60. PMID 15706734
- [Result] Pittler MH, Verster JC, Ernst E. Interventions for preventing or treating alcohol hangover: systematic review of randomised controlled trials. BMJ. 2005 Dec 24;331(7531):1515-8. doi: 10.1136/bmj.331.7531.1515. PMID 16373736
- [Result] Wiese JG, Shlipak MG, Browner WS. The alcohol hangover. Ann Intern Med. 2000 Jun 6;132(11):897-902. doi: 10.7326/0003-4819-132-11-200006060-00008. PMID 10836917
- [Result] Slutske WS, Piasecki TM, Hunt-Carter EE. Development and initial validation of the Hangover Symptoms Scale: prevalence and correlates of Hangover Symptoms in college students. Alcohol Clin Exp Res. 2003 Sep;27(9):1442-50. doi: 10.1097/01.ALC.0000085585.81711.AE. PMID 14506405

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 62 people were enrolled however only 49 were included in the analysis due to not submitting their surveys or did not complete the first day of the study.
Groups:
- NAC First, Then Placebo: Patients receiving NAC after drinking to breathalyzer value 0.1 and then completed the survey in the morning after drinking and then at a later date returned and drank again to BrAC level of 0.1 and received placebo then again completed the survey in the morning
- Placebo First Then NAC Group: Patients receiving placebo after drinking to breathalyzer value 0.1 and then completed the survey in the morning after drinking and then at a later date returned and drank again to BrAC level of 0.1 and received NAC then again completed the survey in the morning
Period: First Intervention
Arm/Group | NAC First, Then Placebo | Placebo First Then NAC Group
Started | 23 | 26
Completed | 23 | 26
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | NAC First, Then Placebo | Placebo First Then NAC Group
Started | 23 | 26
Completed | 23 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants received the 2 interventions - NAC and placebo. The participants completed one intervention on one day and returned to complete the other intervention on a subsequent day.
Arm/Group | All Study Participants
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 49
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Hangover Symptom Scale
Description: In the morning, each participate will fill out a Hangover Symptom Score questionnaire, evaluating each hangover symptom on a 0 - 4 point Hangover Symptom Severity scale. 0 representing "strongly disagree" or "feels like I did not drink last night" to 4 representing "strongly agree" or "I'm so hungover / I'm never drinking again" for each symptom. The symptoms on the Hangover Symptom Scale are: feeling thirsty or dehydrated, feeling more tired than usual, headache, nauseated, vomited, feeling weak, difficulty concentrating, more sensitive to light and sound than usual, sweating more than usual, had trouble sleeping, feeling anxious, feeling depressed, experienced trembling or shaking. The total score could range from 0-52 with 0 being no symptoms of hangover and 52 being the worst symptoms of hangover. This study looked specifically at the overall hangover score, nauseated, feeling weak and headache.
Time Frame: 12 hours or less
Measure: Median (Full Range); unit: units on a scale
Groups:
- NAC Group: Patients receiving NAC after drinking to breathalyzer value 0.1
  N Acetyl Cysteine
- Placebo Group: Patients receiving placebo after drinking to breathalyzer value 0.1
  placebo
Arm/Group | NAC Group | Placebo Group
Number analyzed (Participants) | 49 | 49
units on a scale
  total Hangover symptom score | 10 [0 to 35] | 13 [0 to 38]
  headache | 1 [0 to 4] | 1 [0 to 4]
  nauseated | 0 [0 to 4] | 1 [0 to 4]
  feeling weak | 1 [0 to 4] | 1 [0 to 4]
Statistical Analysis 1: Comparison: NAC Group vs Placebo Group; Test type: Superiority; p = 0.45, Wilcoxon (Mann-Whitney) — p-value calculated for the total hangover scale
Statistical Analysis 2: Comparison: NAC Group vs Placebo Group; Test type: Superiority; p = 0.93, Wilcoxon (Mann-Whitney) — p value calculated for symptom of headache
Statistical Analysis 3: Comparison: NAC Group vs Placebo Group; Test type: Superiority; p = 0.11, Wilcoxon (Mann-Whitney) — p value calculated for symptom of nausea
Statistical Analysis 4: Comparison: NAC Group vs Placebo Group; Test type: Superiority; p = 0.72, Wilcoxon (Mann-Whitney) — p value calculated for symptom of weakness

ADVERSE EVENTS:
Time Frame: 20 hours
Arm/Group | NAC Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 11/49 | 4/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NAC Group (N=49) | Placebo Group (N=49)
gas (Gastrointestinal disorders) | 3 | 0
insomnia (Nervous system disorders) | 1 | 0
bloating (Gastrointestinal disorders) | 1 | 0
acid reflux (Gastrointestinal disorders) | 1 | 0
muscle twitches (Musculoskeletal and connective tissue disorders) | 1 | 0
stomach pain (Gastrointestinal disorders) | 1 | 0
diarrhea (Gastrointestinal disorders) | 1 | 0
headache (Nervous system disorders) | 1 | 3
rash (Skin and subcutaneous tissue disorders) | 1 | 0
vomiting (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes